CLINICAL TRIAL: NCT00531661
Title: CardioMEMS Heart Sensor Allows Monitoring of Pressure to Improve Outcomes in NYHA Class III Heart Failure Patients
Acronym: CHAMPION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CardioMEMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CM-06-04
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TREATMENT Group (Active Comparator): Standard of care HF management plus HF management based upon hemodynamic information obtained from the HF Pressure Measurement System
  Interventions: Device: HF Pressure Measurement System
- CONTROL Group (Placebo Comparator): Standard of care HF management

INTERVENTIONS:
Device: HF Pressure Measurement System — A pressure sensor is intended to be implanted into the pulmonary artery at the time of Swan-Ganz catheterization.
  Arms: TREATMENT Group

SUMMARY:
This is a prospective, multi-center, randomized, single-blind clinical trial conducted in the United States (US). The objective of the study is to evaluate the safety and efficacy of the HF Pressure Measurement System in reducing heart failure (HF) related hospitalizations in a subset of subjects suffering from HF.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HF ≥ 3 months, with either preserved or reduced LVEF
2. Diagnosis of NYHA Class III HF (historical assessment documented at screening visit)
3. Subjects with reduced LVEF must be receiving a beta blocker for 3 months and an ACE-I or ARB for one month unless in the investigator's opinion, the subject is intolerant to beta blockers, ACE-I or ARB. Beta blockers and ACE-I (or ARB) doses should be stable for one month prior to study entry.
4. At least 1 HF hospitalization within 12 months of Screening Visit
5. Subjects with pulmonary artery branch diameter sized between 7mm and 15mm (implanted vessel)

Exclusion Criteria:

1. Subjects with history of recurrent (> 1) pulmonary embolism or deep vein thrombosis
2. Subjects, in the Investigator's opinion, unable to tolerate a right heart catheterization
3. Subjects who have had a major cardiovascular event (e.g., myocardial infarction, stroke) within 2 months of Screening Visit
4. Subjects with Cardiac Resynchronization Device (CRT) implanted ≤ 3 months prior to enrollment
5. Subjects with a Glomerular Filtration Rate (GFR) <25 ml/min who are non-responsive to diuretic therapy or who are on chronic renal dialysis
6. Subjects likely to undergo heart transplantation within 6 months of Screening Visit
7. Subjects with congenital heart disease or mechanical right heart valve(s)
8. Subjects with known coagulation disorders
9. Subjects with a hypersensitivity or allergy to aspirin, and/or clopidogrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2007-09; Primary Completion 2010-05 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Adamson, MD, FACC, Principal Investigator — Oklahoma Heart Hospital; William T Abraham, MD, FACC, Principal Investigator — Ohio State University
Locations (1):
- CardioMEMS Investigational Sites, Nationwide, Georgia, United States

REFERENCES:
- [Derived] Zile MR, Abraham WT, Stevenson LW, Costanzo MR, Angermann CE, Mehra MR, Desai AS, Ducharme A, Johnson N, Henderson J, Lindenfeld J. Relationship Between Remote, Ambulatory Pulmonary Artery Pressures, and All-Cause Mortality in Patients With Chronic Heart Failure. Circ Heart Fail. 2025 Jun;18(6):e012754. doi: 10.1161/CIRCHEARTFAILURE.124.012754. Epub 2025 Apr 14. PMID 40223608
- [Derived] Varma N, Bourge RC, Stevenson LW, Costanzo MR, Shavelle D, Adamson PB, Ginn G, Henderson J, Abraham WT; CHAMPION Investigator Group. Remote Hemodynamic-Guided Therapy of Patients With Recurrent Heart Failure Following Cardiac Resynchronization Therapy. J Am Heart Assoc. 2021 Feb;10(5):e017619. doi: 10.1161/JAHA.120.017619. Epub 2021 Feb 25. PMID 33626889
- [Derived] Givertz MM, Stevenson LW, Costanzo MR, Bourge RC, Bauman JG, Ginn G, Abraham WT; CHAMPION Trial Investigators. Pulmonary Artery Pressure-Guided Management of Patients With Heart Failure and Reduced Ejection Fraction. J Am Coll Cardiol. 2017 Oct 10;70(15):1875-1886. doi: 10.1016/j.jacc.2017.08.010. PMID 28982501
- [Derived] Adamson PB, Abraham WT, Stevenson LW, Desai AS, Lindenfeld J, Bourge RC, Bauman J. Pulmonary Artery Pressure-Guided Heart Failure Management Reduces 30-Day Readmissions. Circ Heart Fail. 2016 Jun;9(6):e002600. doi: 10.1161/CIRCHEARTFAILURE.115.002600. PMID 27220593
- [Derived] Abraham WT, Stevenson LW, Bourge RC, Lindenfeld JA, Bauman JG, Adamson PB; CHAMPION Trial Study Group. Sustained efficacy of pulmonary artery pressure to guide adjustment of chronic heart failure therapy: complete follow-up results from the CHAMPION randomised trial. Lancet. 2016 Jan 30;387(10017):453-61. doi: 10.1016/S0140-6736(15)00723-0. Epub 2015 Nov 9. PMID 26560249
- [Derived] Raina A, Abraham WT, Adamson PB, Bauman J, Benza RL. Limitations of right heart catheterization in the diagnosis and risk stratification of patients with pulmonary hypertension related to left heart disease: insights from a wireless pulmonary artery pressure monitoring system. J Heart Lung Transplant. 2015 Mar;34(3):438-47. doi: 10.1016/j.healun.2015.01.983. Epub 2015 Feb 7. PMID 25813770
- [Derived] Adamson PB, Abraham WT, Bourge RC, Costanzo MR, Hasan A, Yadav C, Henderson J, Cowart P, Stevenson LW. Wireless pulmonary artery pressure monitoring guides management to reduce decompensation in heart failure with preserved ejection fraction. Circ Heart Fail. 2014 Nov;7(6):935-44. doi: 10.1161/CIRCHEARTFAILURE.113.001229. Epub 2014 Oct 6. PMID 25286913
- [Derived] Abraham WT, Adamson PB, Bourge RC, Aaron MF, Costanzo MR, Stevenson LW, Strickland W, Neelagaru S, Raval N, Krueger S, Weiner S, Shavelle D, Jeffries B, Yadav JS; CHAMPION Trial Study Group. Wireless pulmonary artery haemodynamic monitoring in chronic heart failure: a randomised controlled trial. Lancet. 2011 Feb 19;377(9766):658-66. doi: 10.1016/S0140-6736(11)60101-3. PMID 21315441

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: TREATMENT group: standard of care HF management plus HF management based upon hemodynamic information obtained from the HF Pressure Measurement System
- Control: CONTROL group: standard of care HF management
Period: 6 Months
Arm/Group | Treatment | Control
Started | 270 | 280
Completed | 244 | 254
Not Completed | 26 | 26
Period: Study Duration: 15 Months Avg. Follow-up
Arm/Group | Treatment | Control
Started | 244 | 254
Completed | 186 | 197
Not Completed | 58 | 57

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 270 | 280 | 550
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 150 | 155 | 305
  >=65 years | 120 | 125 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (13.0) | 61.8 (12.7) | 61.6 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 75 | 151
  Male | 194 | 205 | 399
Region of Enrollment [Number; unit: participants]
  United States | 270 | 280 | 550

OUTCOME MEASURES:

1. Primary Outcome: Rate of Heart Failure Related (HFR) Hospitalizations
Time Frame: 6 months
Measure: Number; unit: HFR hospitalizations/patient/6 months
Arm/Group | Treatment | Control
Number analyzed (Participants) | 270 | 280
HFR hospitalizations/patient/6 months | 0.32 | 0.44
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.0002, Negative Binomial Regression

2. Primary Outcome: Freedom From a Device/System-related Complication (DSRC).
Description: A DSRC is an adverse event that is, or is possibly, related to the HF Pressure Measurement System and at least one the following:
  * is treated with invasive means (other than intramuscular medication or a right heart catheterization with a Swan-Ganz measurement which is used for diagnostic purposes)
  * results in the death of the subject
  * results in the explant of the device
Time Frame: 6 months
Population: This Safety Endpoint was prespecified as an aggregate analysis of all patients implanted with the device as well as patients where an implant was attempted. Results are not presented as an inter-arm comparison but rather against an objective performance criteria (OPC). This population includes 550 implanted patients + 25 patient attempts.
Measure: Number; unit: cases
Units Other Than Participants: Implantation Cases
Arm/Group | Entire Study Cohort
Number analyzed (Participants) | 550
Number analyzed (Implantation Cases) | 575
cases | 567 [97.3% to 99.4%]
Statistical Analysis 1: Comparison: Entire Study Cohort; Analysis of DSRC was based on the following pre-specified objective performance criteria: the lower limit of the two-sided 95.2% confidence interval on the freedom from DSRC rate for all implantation cases was at least 80%. The statistical hypotheses were: Null: (Freedom from device / system-related complications) ≤ 80% Alternative: (Freedom from device / system-related complications) > 80%; Test type: Superiority or Other; p < 0.0001, exact test of binomial proportions; P-value from exact test of binomial proportions compared proportion of all implantation cases free from DSRC to OPC of 0.80

3. Primary Outcome: Freedom From Pressure Sensor Failure
Description: A pressure sensor failure occurs when the sensor malfunctions to the point that no readings can be obtained from it after all attempts are exhausted including troubleshooting the system to rule out any problems with the electronic components.
Time Frame: 6 months
Population: This Safety Endpoint was prespecified as an aggregate analysis of all patients implanted with the device. Results are not presented as an inter-arm comparison but rather against an objective performance criteria (OPC).
Measure: Number; unit: participants
Arm/Group | Entire Randomized Study Cohort
Number analyzed (Participants) | 550
participants | 550
Statistical Analysis 1: Comparison: Entire Randomized Study Cohort; Analysis of sensor failures was based on the following pre-specified objective performance criteria: the lower limit of the two-sided 95.2% confidence interval on the freedom from pressure sensor failure rate for all patients implanted was at least 90%. The statistical hypotheses were: Null: (Freedom from device / system-related complications) ≤ 90% Alternative: (Freedom from device / system-related complications) > 90%; Test type: Superiority or Other; p < 0.0001, exact test of binomial proportions; P-value from exact test of binomial proportions compared proportion of all implanted patients free from pressure sensor failure to OPC of 0.90

4. Secondary Outcome: Change From Baseline in Pulmonary Artery Mean Pressure
Description: Change from baseline in pulmonary artery mean pressure was calculated using an area under the curve (AUC) methodology. All patients were instructed to take daily home readings for 180 days. By patient, a baseline average for the first 7 days of home readings was calculated. The difference between baseline and each daily reading was then determined and a corresponding daily AUC value was calculated. Finally, all daily AUC values were summed over the entire 180 day period resulting in a total AUC per patient. These data were aggregated for each randomization group and then compared. The unit of measure is mmHg x Days.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg * days
Arm/Group | Treatment | Control
Number analyzed (Participants) | 270 | 280
mmHg * days | -155.7 (1088.0) | 33.1 (951.7)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.0077, ANCOVA

5. Secondary Outcome: Proportion of Patients Hospitalized for Heart Failure
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 270 | 280
participants | 55 | 80
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.0292, Fisher Exact

6. Secondary Outcome: Days Alive Outside of the Hospital
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment | Control
Number analyzed (Participants) | 270 | 280
days | 174.4 (31.1) | 172.1 (37.8)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.0280, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Quality of Life - Minnesota Living With Heart Failure Questionnaire (MLHFQ)
Description: THe MLHFQ is patient self-assessment of how heart failure affects his or her daily life. To measure the effects of symptoms, functional limitations, psychological distress on an individual's quality of life, the MLHFQ questionnaire asks each person to indicate using a 6-point, zero to five, Likert scale how much each of 21 facets prevented them from living as they desired. Total scores are provided as sums. The total score scale range is 0 - 105. A lower total score is indicative of better quality of life.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 270 | 280
units on a scale | 45.2 (26.4) | 50.6 (24.8)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.0236, t-test, 2 sided

8. Other Pre Specified Outcome: Rate of HFR Hospitalizations
Time Frame: Study duration: average patient follow-up of 15 months
Measure: Number; unit: HFR hospitalizations/patient-year
Arm/Group | Treatment | Control
Number analyzed (Participants) | 270 | 280
HFR hospitalizations/patient-year | 0.46 | 0.73
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p < 0.0001, Negative Binomial Regression

9. Other Pre Specified Outcome: Freedom From a Device/System-related Complication (DSRC)
Time Frame: Study duration: average patient follow-up of 15 months
Measure: Number; unit: participants
Groups:
- Full Duration Study Cohort: Safety endpoint evaluated for all patients having follow-up after the 6-month primary period.
Arm/Group | Full Duration Study Cohort
Number analyzed (Participants) | 498
participants | 498
Statistical Analysis 1: Comparison: Full Duration Study Cohort; Analysis of DSRC was based on the following pre-specified objective performance criteria: the lower limit of the two-sided 95.2% confidence interval on the freedom from DSRC rate for all implanted patients was at least 80%. The statistical hypotheses were: Null: (Freedom from device / system-related complications) ≤ 80% Alternative: (Freedom from device / system-related complications) > 80%; Test type: Superiority or Other; p < 0.0001, exact test of binomial proportions; P-value from exact test of binomial proportions compared proportion of all implanted patients free from DSRC to OPC of 0.80

10. Other Pre Specified Outcome: Freedom From Pressure Sensor Failure
Time Frame: Study duration: average patient follow-up of 15 months
Measure: Number; unit: participants
Arm/Group | Full Duration Study Cohort
Number analyzed (Participants) | 498
participants | 498
Statistical Analysis 1: Comparison: Full Duration Study Cohort; Analysis of sensor failures was based on the following pre-specified objective performance criteria: the lower limit of the two-sided 95.2% confidence interval on the freedom from pressure sensor failure rate for all implanted patients was at least 90%. The statistical hypotheses were: Null: (Freedom from device / system-related complications) ≤ 90% Alternative: (Freedom from device / system-related complications) > 90%; Test type: Superiority or Other; p < 0.0001, exact test of binomial proportions; [statistical method as in outcome 3, analysis 1]

ADVERSE EVENTS:
Arm/Group | Treatment | Control
Serious Adverse Events (participants affected / at risk) | 121/270 | 155/280
Other Adverse Events (participants affected / at risk) | 175/270 | 174/280
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=270) | Control (N=280)
Cardiac Disorders (Cardiac disorders) | 76 (144) | 101 (187)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 22 (26) | 25 (31)
infections (Infections and infestations) | 22 (27) | 22 (24)
vascular (Vascular disorders) | 17 (21) | 15 (16)
renal and urinary (Renal and urinary disorders) | 19 (19) | 12 (13)
metabolism and nutrition (Metabolism and nutrition disorders) | 14 (16) | 12 (13)
nervous system (Nervous system disorders) | 12 (16) | 14 (20)
gastrointestinal (Gastrointestinal disorders) | 12 (18) | 12 (19)
general disorders (General disorders) | 9 (10) | 12 (15)
surgical (Surgical and medical procedures) | 10 (11) | 11 (13)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=270) | Control (N=280)
respiratory (Respiratory, thoracic and mediastinal disorders) | 42 (51) | 44 (62)
cardiac (Cardiac disorders) | 47 (73) | 38 (58)
infections (Infections and infestations) | 38 (50) | 46 (56)
gastrointestinal (Gastrointestinal disorders) | 42 (61) | 34 (49)
metabolism and nutrition (Metabolism and nutrition disorders) | 43 (57) | 29 (33)
nervous system (Nervous system disorders) | 38 (47) | 24 (32)
general disorders (General disorders) | 35 (44) | 24 (30)
musculoskeletal (Musculoskeletal and connective tissue disorders) | 29 (34) | 27 (33)
renal and urinary (Renal and urinary disorders) | 25 (33) | 21 (22)
vascular (Vascular disorders) | 24 (30) | 21 (23)
investigations (Investigations) | 19 (25) | 16 (19)
blood and lymphatic system (Blood and lymphatic system disorders) | 17 (20) | 13 (16)
psychiatric (Psychiatric disorders) | 17 (19) | 12 (14)
skin and subcutaneous tissue (Skin and subcutaneous tissue disorders) | 15 (15) | 13 (15)
injury (Injury, poisoning and procedural complications) | 15 (17) | 12 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No